CLINICAL TRIAL: NCT05508698
Title: Pre-visit Questionnaire to Increase Influenza Vaccinations
Brief Title: Flu Shot Pre-visit Questionnaire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Christopher F Chabris, PhD, Professor, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0419
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Influenza
Keywords: Vaccination; Health Promotion; Health Behavior; Reminder Systems; Economics, Behavioral
MeSH Terms: conditions — Influenza, Human; Health Behavior; Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient-participants will not be explicitly told about the different arms, although clinician-participants will see the different arms and may notice these differences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive Control (No Intervention): No change to the standard of care for flu vaccines
- Pre-visit Questionnaire (Experimental): One-item questionnaire in online patient portal and additional information in the flu shot alert
  Interventions: Behavioral: Precommitment Nudge; Behavioral: Salience

INTERVENTIONS:
Behavioral: Precommitment Nudge — Ask participants to commit to a decision about getting a flu shot
  Arms: Pre-visit Questionnaire
Behavioral: Salience — Additional text and icon in the flu shot alert makes the pre-visit questionnaire response salient to the clinician, which could facilitate action or further discussion with the patient
  Arms: Pre-visit Questionnaire

SUMMARY:
The purpose of this study is to assess, prospectively, the effect on flu vaccination rates of a pre-visit questionnaire that asks patients to indicate their preferences for a flu shot. Responses to the questionnaire will also be shown to clinicians via additional text in an existing flu shot alert. The investigators hypothesize that the pre-visit questionnaire will lead to increased flu vaccination compared with standard practices.

DETAILED DESCRIPTION:
The CDC (Centers for Disease Control and Prevention) recommends a flu vaccination to everyone aged 6+ months, with rare exception; almost anyone can benefit from the vaccine, which can reduce illnesses, missed work, hospitalizations, and death. One barrier to vaccination is a lack of "cues to action," which could be overcome by asking patients for a pre-visit commitment to get a flu shot and additional reminders for the clinician to act on this commitment.

Eligible patients will be randomized to either receive or not receive a one-item, pre-visit questionnaire about the flu shot (that will show responses to clinicians in an existing flu shot alert).

ELIGIBILITY:
Patient Inclusion Criteria:

* On a list of active Geisinger patients (all patients on this list attended at least one primary care appointment at Geisinger between 10/1/2008 and 4/13/2022, and either had a Geisinger primary care provider assigned as of April 2022, or were in the Electronic Health Record [EHR] since at least September 2021 and had at least one encounter in 2020-2022)
* Has an upcoming flu shot-eligible outpatient visit with a provider
* Has activated Geisinger's patient portal
* Has not yet received a flu vaccine at the time the questionnaire became available, according to the EHR

Clinician Inclusion Criteria

* Any Geisinger clinician who sees patient-participants in our study for a flu shot-eligible outpatient visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230962 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-04-08 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Count of patients with a flu vaccination | Up to 21 days
  Patient received a flu vaccine (yes/no) between the day questionnaires became available for the patient's first scheduled flu-shot-eligible appointment and 7 days following the appointment. Questionnaires were available 14 days prior to the appointment date for appointments scheduled at least 14 days in advance. Questionnaires were available on the day the appointment was scheduled for appointments scheduled less than 14 days in advance.
  Note that control patients did not receive a flu shot questionnaire, but they may have received other questionnaires from the health system 14 days before their appointment. We will conduct subgroup analyses for people who had responded to MyGeisinger pre-visit messages in the previous year and those who did not.

OTHER OUTCOMES:
Count of patients with a high confidence flu diagnosis | Up to 8 months
  Patient received a flu diagnosis via a positive polymerase chain reaction [PCR]/antigen/molecular test (yes/no) during the 2022-23 flu season (from the patient's appointment date through April 30, 2023)
Count of patients with a "likely flu" diagnosis | Up to 8 months
  Received a "high confidence flu" diagnosis (with positive polymerase chain reaction [PCR]/antigen/molecular test) and/or "likely flu" diagnosis (as assessed via International Classification of Disease [ICD] codes or Tamiflu administration or positive PCR/antigen/molecular test) (yes/no) during the 2022-23 flu season (from the patient's appointment date through April 30, 2023)
  Note that "likely flu" is a superset of the "high confidence flu" diagnoses
Count of patients with flu complications | Up to 8 months
  Diagnosed with flu-related complications (yes/no) during the 2022-23 flu season (from the patient's appointment date through April 30, 2023)
ER visits | Up to 11 months
  Number of ER visits from the patient's message appointment date through July 31, 2023
Hospitalizations | Up to 11 months
  Number of hospitalizations from the patient's message appointment date through July 31, 2023
COVID-19 vaccination rates | Up to 8 months
  Received at least one COVID-19 vaccination (yes/no) during the 2022-23 flu season (from the patient's appointment date through April 30, 2023)
Count of patients with a flu vaccination during the 2022-2023 season | Up to 8 months
  Patient receives a flu vaccine (yes/no) during the 2022-23 flu season (from the patient's appointment date through April 30, 2023)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher F Chabris, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: By the paper's online publication date. Data will remain available for as long as the Open Science Framework hosts it.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT05508698/Prot_SAP_001.pdf